CLINICAL TRIAL: NCT06235359
Title: Is Intercostal Tube Enough in Management of Empyema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Abdelfatah mahmoud, physician, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: empyema
Record Dates: First submitted 2023-10-11; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Empyema
MeSH Terms: conditions — Empyema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intercostal tube (Other): A chest tube is a hollow, flexible tube placed into the chest. It acts as a drain.
  Chest tubes drain blood, fluid, or air from around your lungs, heart, or esophagus.
  The tube around your lung is placed between your ribs and into the space between the inner lining and the outer lining of your chest cavity. This is called the pleural space. It allows your lungs to fully expand.
  Interventions: Device: intercostal tube

INTERVENTIONS:
Device: intercostal tube — A chest tube is a hollow, flexible tube placed into the chest. It acts as a drain.
  Chest tubes drain blood, fluid, or air from around your lungs, heart, or esophagus.
  The tube around your lung is placed between your ribs and into the space between the inner lining and the outer lining of your chest cavity. This is called the pleural space. It allows your lungs to fully expand.

SUMMARY:
Is intercostal tube enough in management of empyema ?

DETAILED DESCRIPTION:
Empyema refers to presence of pus in the pleural space -Causes Primary: bacterial Pneumonia (staph aureus, strept pneumonia , H.influenza) , TB

Secondry :

PostTraumati postoperative :open heart , esophageal, mediastinum , lung rupture of lung absess

-pathophysiology and stages During an inflammatory process such as pneumonia, there is an increase in fluid production in the pleural cavity known as the exudate stage. As the disease progresses microorganisms, usually bacteria, can colonize the fluid and generated an empyema. This fluid is characterized by elevated lactate dehydrogenase, proteins, neutrophils, and dead cells. Macroscopically is a thick opaque fluid found in the fibrinopurulent stage. After the resolution of the infection and as a consequence of the inflammation, there is a process of fibrosis that can lead to restriction of the lung parenchyma which is stage of chronic organization

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to Assuit university Hospital and diagnosed with empyema

Exclusion Criteria:

* Patient diagnosed with Post-operative empyema
* Patient diagnosed with post traumatic empyema
* Patient diagnosed with Bronchopleural fistula
* Patient diagnosed with TB

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To find best way to drain the pus in the pleural space | baseline
  To find best way to drain the pus in the pleural space

REFERENCES:
- [Background] Ali I, Unruh H. Management of empyema thoracis. Ann Thorac Surg. 1990 Sep;50(3):355-9. doi: 10.1016/0003-4975(90)90474-k. PMID 2400254